CLINICAL TRIAL: NCT01449786
Title: Sublingual Immunotherapy of Birch Pollen Associated Apple Allergy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Austrian Science Fund (FWF) (Other)
Responsible Party: Principal Investigator, Tamar Kinaciyan, MD, MD, Ass.Prof., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TK01/2011
Record Dates: First submitted 2011-10-05; First posted 2011-10-10 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Birch Pollen Related Apple Allergy; Birch Pollen Allergy
Keywords: Mal d 1, Bet v 1, sublingual immunotherapy,

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- treatment with rMal d 1 (Experimental): these apple and birch pollen allergic patients are treated with daily sublingual application of 25µg recombinant Major apple allergen, Mal d 1 during 4 months
  Interventions: Drug: rMal d 1
- treatment with rBet v 1 (Active Comparator): These apple and birch pollen allergic patients are treated with daily sublingual application of 25µg recombinant Major birch pollen allergen,Bet v 1 during 4 months
  Interventions: Drug: rBet v 1
- treatment with placebo drops (Placebo Comparator): These apple and birch pollen allergic patients are treated daily with placebo applied sublingually during 4 months
  Interventions: Other: placebo drops

INTERVENTIONS:
Drug: rMal d 1 — 25 µg daily as sublingually administered drops, 16 weeks
  Arms: treatment with rMal d 1
Drug: rBet v 1 — 25 µg daily administered sublingually as drops over 16 weeks
  Arms: treatment with rBet v 1
Other: placebo drops — 25 µg of placebo Drops daily administered sublingually over 16 weeks
  Arms: treatment with placebo drops

SUMMARY:
More than 70% of birch pollen allergic patients suffer from allergic reactions to certain foods, e.g. stone fruits, hazelnut and some vegetables. However, specific immunotherapy (SIT) with birch pollen extract is not effective for the treatment of associated food allergy in a substantial number of patients. Based on our previous clinical and immunological investigations of birch pollen related food allergy (BPRFA) the investigators hypothesize that for effective SIT of this abundant food allergy the disease-eliciting food allergens should be employed. To prove this concept, the investigators aim to sublingually administer the major apple allergen, Mal d 1, to birch pollen-allergic patients with concomitant apple allergy and evaluate clinical and immunological effects of this treatment. The investigators choose Mal d 1 as model food allergen because (i) its cross-reactivity with Bet v 1 has been well characterized,(ii) apple is the most frequent trigger for BPRFA and (iii) recombinant(r)Mal d 1 was well tolerated after sublingual administration to 20 birch pollen-allergic patients in a previous study. Sublingual administration of a defined concentration of GMP-rMal d 1 will be compared with equal doses of GMP-rBet v 1 as a positive control and placebo-treatment. Clinical parameters will include skin prick tests (SPT) and objective and subjective assessment of apple and birch pollen-induced allergic symptoms. Immunological parameters will comprise the analysis of antibody and T cell responses to Mal d 1 and Bet v 1 as well as the evaluation of basophil activation.

The proposed pilot study will be a first investigation of the concept to specifically treat BPRFA with the involved food allergens and thus, represents an important step in the development of an efficient and safe therapy in the future.

ELIGIBILITY:
Inclusion Criteria:

* otherwise healthy persons between 18 und 50 years of age;
* positive history of rhinoconjunctivitis to birch pollen
* oral allergy syndrome(OAS) to apple
* positive skin prick test (SPT) reaction to birch pollen and apple
* specific IgE for Bet v 1 and Mal d 1

Exclusion Criteria:

* Exclusion criteria
* Persons who due to their physical or mental state are not able to provide informed consent.
* Persons with underlying illnesses such as severe cardiopulmonary, malignant and/or autoimmune diseases
* Persons suffering from Hyper-IgE syndrome
* Persons receiving SIT during the past 5 years
* persons suffering from severe allergic reactions to apple such as generalized urticaria, asthma and/or anaphylaxis
* persons suffering from severe bronchial asthma to birch pollen
* persons suffering from pathological alterations of the lips and oral mucosa
* persons who are prescribed a treatment with immune-suppressive drugs, anti-histamines, leukotriene-antagonists or psychotropic drugs with anti-histaminic effects
* persons using ß-blockers
* Pregnant woman

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03-14 (Actual); Primary Completion 2014-02-28 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
allergen concentration to induce allergic reactions in the oral cavity as a measure of efficacy (oral provocation test) | 1 year
  To measure the clinical effects on apple-induced OAS, open food challenges (OFC) with every 30 minutes increasing doses of GMP-rMal d 1 will be performed before and after the treatment period.

SECONDARY OUTCOMES:
T cell proliferation and cytokine production as a measure of tolerance induction | 1 year
  PBMC isolated from heparinised blood before, during and after sublingual administration of the treatment will be stimulated with titrated concentrations of rMal d 1 and rBet v 1, respectively. Proliferative and cytokine responses will be determined.
allergen specific antibody response | 1
  measurement of IgE, IgG and IgA antibodies specific for Bet v 1 and Mal d 1

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Bohle, PhD, Prof., Principal Investigator — Medical University of Vienna; Tamar Kinaciyan, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No